CLINICAL TRIAL: NCT06194760
Title: Evaluation of Vitrectomy With ILM Peeling in Myopic Macular Hole With Only Posterior Retinal Detachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Tharwat, Principal Investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vitrectomy with ILM peeling
Record Dates: First submitted 2023-12-23; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- myopic eyes with macular hole and only posterior retinal detachment (Other)
  Interventions: Procedure: Vitrectomy with ILM peeling

INTERVENTIONS:
Procedure: Vitrectomy with ILM peeling — Vitrectomy with traditional internal limiting membrane (ILM) peeling technique is regarded as the gold standard treatment for MH; it works by completely relieving of the traction of the macula and increasing the flexibility of the retina

SUMMARY:
Retinal detachment (RD) resulting from the macular hole (MH), also known as MH-induced RD (MHRD), most commonly occurs in eyes with high myopia and results in irreversible visual disorders. Although ILM peeling for MHRD reportedly achieves a high retinal reattachment rate that ranges from 70% to 100%, the MH closure rate is relatively low, ranging from 10% to 70%.

ELIGIBILITY:
Inclusion Criteria:

* patients with high myopia (a spherical equivalent refractive error of at least -6.0 diopters (D) and an axial length of at least 26.5 mm).
* Macular hole and only posterior retinal detachment

Exclusion Criteria:

* Other causes of RD
* Patients with a history of trauma, choroidal neovascularization, coexistence with a peripheral retinal break or proliferative vitreoretinopathy
* History of any vitreoretinal surgery prior to MHRD and less than 36 months of follow-up after the surgery

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Closure of macular hole | 6 months post operative
  It is a subjective outcome measured by Optical coherence tomography and by clinical slit lamb examination
BCVA | baseline
  It is a measure of the visual acuity, which will be measured by LogMar
BCVA | 6 months postoperative
  It is a measure of the visual acuity, which will be measured by LogMar
BCVA | 12 months postoperative
  It is a measure of the visual acuity, which will be measured by LogMar

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No